CLINICAL TRIAL: NCT01409096
Title: A Randomized, Double Blind, Placebo-controlled Trial of Pregnenolone for Bipolar Depression
Brief Title: Study Using Pregnenolone to Treat Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Sherwood Brown, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 122009-069
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Bipolar Disorder; Major Depressive Disorder
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major | interventions — Pregnenolone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregnenolone (Active Comparator): This arm will be given 50mg Pregnenolone twice per day for 2 weeks, then 150mg Pregnenolone twice per day for 2 weeks, then 250mg Pregnenolone twice per day for 8 weeks.
  Interventions: Drug: Pregnenolone
- Placebo (Placebo Comparator): The arm will be given placebo that matches the Pregnenolone at the same frequency as the Pregnenolone for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone — Pregnenolone is a naturally occurring neurosteroid that is synthesized from cholesterol in the adrenal glands and central nervous system.
  Other Names: 3β-hydroxypregn-5-en-20-one
  Arms: Pregnenolone
Drug: Placebo — Inactive ingredient matching the active medication in appearance.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Primary purpose of this study is to determine if pregnenolone supplementation is associated with greater improvement in depressive symptoms of patients with bipolar disorder. Also the study will explore possibilities of improving anxiety and manic symptoms as well as the patient's cognition.

DETAILED DESCRIPTION:
Determine if pregnenolone supplementation is associated with greater improvement in depressive symptoms than placebo in persons with Bipolar Depression (BPD), depressed phase. In our pilot study, pregnenolone showed a strong signal on depression scores.

Secondary

1. Determine if pregnenolone supplementation is associated with greater improvement in anxiety symptoms in persons with BPD, depressed phase. Data from prior studies suggests that pregnenolone may decrease symptoms of anxiety. Anxiety is a common and clinically important feature of BPD. Therefore, we will examine anxiety symptoms in this trial.
2. Determine if pregnenolone supplementation is associated with improvement in manic symptoms as compared to placebo in persons with BPD, depressed phase. Our pilot study suggested that pregnenolone may be associated with improvement in manic symptoms. Although the current study targets bipolar depression we will also examine manic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women of all races age 18-75 years
* Diagnosis of bipolar I, II or not otherwise specified (NOS) disorders currently meeting criteria for a major depressive episode
* English speaking

Exclusion Criteria:

* Active suicidal ideation with plan and intent
* Treatment resistant depression
* Vulnerable population (i.e. pregnant, cognitively impaired, incarcerated)
* Severe or life threatening medical condition
* History of allergic reaction or side effects with prior pregnenolone use
* Current substance use disorder defined as meeting criteria for abuse or dependence based on the Structured Clinical Interview for the Diagnostic and Statistical Manual (DSM)(SCID) interview and self-reported use within the past 3 months or a positive baseline urine drug screen
* Removal or addition of concomitant psychiatric medications within 10 days prior to randomization
* Current Warfarin therapy
* Current use of oral contraceptives
* Current hormone replacement therapy
* History of heart disease or arrhythmias
* Current (past 7 days) systemic

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edson S Brown, MD/PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregnenolone | Placebo
Started | 40 | 40
Completed | 38 | 35
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnenolone | Placebo | Total
Number analyzed (Participants) | 38 | 35 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (8.5) | 44.1 (10.4) | 43.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 24 | 40
  Male | 22 | 11 | 33
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 18 | 15 | 33
  Caucasian | 18 | 16 | 34
  Hispanic | 2 | 4 | 6
Bipolar Diagnosis [Number; unit: participants] — Participants were graded clinically by using the Diagnostic and Statistical Manual of Mental Disorders (DSM) guidelines for criteria from a structured clinical interview.
  participants
    Bipolar I | 16 | 15 | 31
    Bipolar II | 21 | 17 | 38
    Bipolar Not Otherwise Specified | 1 | 3 | 4
Age of onset of mood symptoms [Mean (Standard Deviation); unit: years] | 26.4 (9.0) | 26.7 (7.3) | 26.7 (8.22)
Concomitant Medications: Lithium [Number; unit: participants]
  Lithium | 5 | 4 | 9
  No Lithium | 33 | 31 | 64
Concomitant Medications: Anticonvulsant [Number; unit: participants]
  Anticonvulsants | 10 | 10 | 20
  No anticonvulsants | 28 | 25 | 53
Concomitant Medications: Antidepressant [Number; unit: participants]
  Antidepressants | 21 | 22 | 43
  No antidepressants | 17 | 13 | 30
Concomitant Medications: Antipsychotic [Number; unit: participants]
  Antipsychotic | 17 | 18 | 35
  No antipsychotic | 21 | 17 | 38
Concomitant Medications: Sedative/hypnotic/anxiolytic [Number; unit: participants]
  Sedative/hypnotic/anxiolytic | 16 | 20 | 36
  No Sedative/hypnotic/anxiolytic | 22 | 15 | 37
Concomitant medications: Stimulant [Number; unit: participants]
  Stimulant | 0 | 1 | 1
  No stimulant | 38 | 34 | 72
Concomitant medications: None [Number; unit: participants]
  No concomitant medications | 7 | 6 | 13
  Concomitant medication | 31 | 29 | 60
Hamilton Rating Scale for Depression (HRSD) [Mean (Standard Deviation); unit: units on a scale] — Minimum: 0 Maximum: 50 Better outcome: lower Normal= 7 or less
  units on a scale | 21.3 (4.0) | 23.5 (4.6) | 22.4 (4.3)
Inventory of Depressive Symtomatology-Self Report (IDS-SR) [Mean (Standard Deviation); unit: units on a scale] — Minimum: 0 Maximum: 84 Better outcome: Lower Normal: 7 or less
  units on a scale | 38.0 (14.5) | 47.5 (14.5) | 42.7 (15.2)
Young Mania Rating Scale (YMRS) [Mean (Standard Deviation); unit: units on a scale] — Minimum: 0 Maximum: 60 Better outcome: lower
  units on a scale | 10.1 (4.7) | 10.4 (4.3) | 10.1 (4.3)
Hamilton Rating Scale for Anxiety (HRSA) [Mean (Standard Deviation); unit: units on a scale] — Minimum: 0 Maximum: 56 Better outcome: lower
  units on a scale | 19.4 (9.8) | 22.8 (8.1) | 21.1 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: The 17-item Hamilton Rating Scale for Depression (HRSD17)
Description: The HRSD is an observer-rated measure of depressive symptomatology.
  Minimum: 0; Maximum: 50; Better outcome: lower score; Normal score: 7 or less.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 38 | 35
units on a scale | 9.18 (1.41) | 9.41 (1.35)
Statistical Analysis 1: Comparison: Pregnenolone vs Placebo; Baseline HRSD scores used as covariate; Test type: Superiority or Other; p = 0.9084, ANCOVA

2. Secondary Outcome: Inventory of Depressive Symptomatology-Self Report (IDS-SR)
Description: IDS-SR is a self reported 30 item assessment to diagnose a major depressive episode.
  Score:
  Minimum: 0 Maximum: 84 Lower score associated with better outcome
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 38 | 35
units on a scale | 15.78 (2.64) | 18.23 (2.54)
Statistical Analysis 1: Comparison: Pregnenolone vs Placebo; Baseline IDS-SR used as a covariate; Test type: Superiority or Other; p = 0.5187, ANCOVA

3. Secondary Outcome: Young Mania Rating Scale (YMRS)
Description: This is an 11-item, observer rated measure of the severity of manic symptoms on a 5 point scale. The total score indicates overall severity of mania with a minimum of zero (indicating normalcy) and a maximum of 60 (indicating very severe).
  Score:
  Minimum: 0 Maximum: 60 Lower score associated with better outcome
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 38 | 35
units on a scale | 5.84 (1.09) | 6.63 (1.05)
Statistical Analysis 1: Comparison: Pregnenolone vs Placebo; Baseline YMRS used as a covariate; Test type: Superiority or Other; p = 0.6060, ANOVA

4. Secondary Outcome: Hamilton Rating Scale for Anxiety (HRSA)
Description: The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety).
  Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where less than 17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 38 | 35
units on a scale | 8.80 (1.63) | 10.32 (1.57)
Statistical Analysis 1: Comparison: Pregnenolone vs Placebo; Baseline HRSA used as a covariate; Test type: Superiority or Other; p = 0.5110, ANCOVA

ADVERSE EVENTS:
Arm/Group | Pregnenolone | Placebo
Serious Adverse Events (participants affected / at risk) | 4/38 | 3/35
Other Adverse Events (participants affected / at risk) | 0/38 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregnenolone (N=38) | Placebo (N=35)
Corneal ulceration (Eye disorders) | 1 (1) | 0 (0)
Skin abscess followed by allergic reaction to antibiotic used to treat it (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Injuries secondary to motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Sample size; treatment groups not well matched on gender or depressive symptom scores

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No